CLINICAL TRIAL: NCT07050485
Title: Postbiotics for Mitigation of Postoperative Dysbiosis in Gastrointestinal Cancer Surgery: A Randomized, Single-blinded, Placebo-controlled Trial (REPOT)
Brief Title: Postbiotics for Mitigation of Postoperative Dysbiosis in Gastrointestinal Cancer Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPOT
Record Dates: First submitted 2025-06-20; First posted 2025-07-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Treatment group will receive PoZibio at a dose of 1 gummy once daily for 7 days prior to surgery and 90 days post surgery. Pozibio will be administered as a chewable gummy formulation, to be taken orally at approximately the same time each day.
  Interventions: Dietary Supplement: PoZibio
- Control Group (Placebo Comparator): Control group will receive an inert placebo gummy, matched in appearance, taste, texture, and packaging to Pozibio®. The placebo will also be taken once daily for 7 days prior to surgery and 90 days post surgery, following the same schedule as the Test group.
  Interventions: Dietary Supplement: Inert placebo

INTERVENTIONS:
Dietary Supplement: PoZibio — 1 gummy once daily
  Arms: Treatment Group
Dietary Supplement: Inert placebo — 1 gummy once daily
  Arms: Control Group

SUMMARY:
To measure the efficacy of postbiotic supplements in mitigating the gut dysbiosis induced by colon cancer surgery. Efficacy in mitigating dysbiosis will be measured by the change in fecal Shannon Diversity Index (SDI) within patients from the baseline sample to various postoperative timepoints. Mean change in SDI from baseline will be compared between groups at 2 weeks postoperative

DETAILED DESCRIPTION:
This is a randomized, single-blinded study designed to assess the efficacy of postbiotic supplements in mitigating gut dysbiosis induced during the perioperative period of laparoscopic colon cancer surgery. Eligible participants, who are scheduled to undergo laparoscopic colon cancer surgery according to standard clinical procedures, will be enrolled following informed consent. Once consent is obtained, participants who meet the eligibility criteria will be randomly assigned in a 1:1 ratio to either the Treatment group or the Control group. Both groups will take 1 gummy once daily ≥ 7 days prior to surgery and 90 days post surgery. Stool samples will be collected at five timepoints, along with a portion of the tumor tissue resected at surgery. The collected samples will be compared between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Recently diagnosed with nonmetastatic GI cancer, including but not limited to small bowel, colon, rectal, pancreatic, gastric, or hepatic malignancies, and scheduled for an elective laparoscopic curative-intent surgical resection in 6 days
2. Able and willing to provide informed consent
3. Age 18 years and above

Exclusion Criteria:

1. Exposed to antibiotics in the 3 months prior to enrollment (per patient-provided history)
2. Unlikely to comply with protocol as determined by Investigator
3. Prior use of any investigational drug in the preceding 6 months prior to enrollment
4. Patients with inflammatory bowel disease
5. Inability to give consent due to a mental condition that makes the participant unable to understand the study's nature, scope, and possible consequences.
6. Emergency surgery
7. Prisoners
8. Known allergy or intolerance to ingredients commonly used in gummy supplements (e.g., gelatin, corn syrup, artificial colors, or natural flavors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in fecal Shannon Diversity Index (SDI) | Baseline, 2 weeks after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at 2 weeks after surgery and baseline between two groups

SECONDARY OUTCOMES:
Change in fecal SDI | Baseline, 3 months after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at after surgery and baseline between two groups
Change in fecal SDI | Baseline, 12 months after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at after surgery and baseline between two groups
Change in fecal SDI | 1 week before surgery, 2 weeks after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at after surgery and baseline between two groups
Change in fecal SDI | 1 week before surgery, 3 months after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at after surgery and baseline between two groups
Change in fecal SDI | 1 week before surgery, 12 months after surgery
  The SDI is a number that reflects both the variety and balance of bacteria in the sample. A higher number means a more diverse bacterial community. Change in fecal SDI is difference at after surgery and baseline between two groups
Change in pathogenic overgrowth in fecal microbiota | Baseline, 2 weeks after surgery
  The relative mean abundance of specific potential pathogenic bacterial species will be measured in fecal samples. An increase in relative abundance may indicate potential overgrowth. Change in pathogenic overgrowth is difference between after surgery and baseline between groups
Change in pathogenic overgrowth in fecal microbiota | 3 months after surgery
  The relative mean abundance of specific potential pathogenic bacterial species will be measured in fecal samples. An increase in relative abundance may indicate potential overgrowth. Change in pathogenic overgrowth is difference between after surgery and baseline between groups
Change in pathogenic overgrowth in fecal microbiota | 12 months after surgery.
  The relative mean abundance of specific potential pathogenic bacterial species will be measured in fecal samples. An increase in relative abundance may indicate potential overgrowth. Change in pathogenic overgrowth is difference between after surgery and baseline between groups
Digestion-associated quality of life questionnaire (DQLQ) scores | Baseline
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. This is compared between groups.
DQLQ scores | 1 week before surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. This is compared between groups.
DQLQ scores | 2 weeks after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. This is compared between groups.
DQLQ scores | 3 months after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. This is compared between groups.
DQLQ scores | 12 months after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. This is compared between groups.
Change in DQLQ scores | Baseline, 2 weeks after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. Change in DQLQ score is difference between after surgery and before surgery between groups.
Change in DQLQ scores | 3 months after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. Change in DQLQ score is difference between after surgery and before surgery between groups.
Change in DQLQ scores | 12 months after surgery
  DQLQ includes 9 statements that assess how often digestive events and experiences affected the physical and mental aspects of quality of life over the past 7 days. The score ranges from 0-9. A higher score indicates a lower (worse) digestion-associated quality of life. Change in DQLQ score is difference between after surgery and before surgery between groups.
Beta diversity of intratumoral microbiomes | Day 0
  Comparison of microbial community composition between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jacobson, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh CK, Huh JW, Lee YJ, Choi MS, Pyo DH, Lee SC, Park SM, Shin JK, Park YA, Cho YB, Yun SH, Kim HC, Lee WY. Long-term Oncologic Outcome of Postoperative Complications After Colorectal Cancer Surgery. Ann Coloproctol. 2020 Aug;36(4):273-280. doi: 10.3393/ac.2019.10.15. Epub 2019 Nov 13. PMID 32054256
- [Result] Nors J, Gotschalck KA, Erichsen R, Andersen CL. Incidence of late recurrence and second primary cancers 5-10 years after non-metastatic colorectal cancer. Int J Cancer. 2024 Jun 1;154(11):1890-1899. doi: 10.1002/ijc.34871. Epub 2024 Feb 7. PMID 38323453
- [Result] Song M, Chan AT, Sun J. Influence of the Gut Microbiome, Diet, and Environment on Risk of Colorectal Cancer. Gastroenterology. 2020 Jan;158(2):322-340. doi: 10.1053/j.gastro.2019.06.048. Epub 2019 Oct 3. PMID 31586566
- [Result] Shogan BD, Smith DP, Christley S, Gilbert JA, Zaborina O, Alverdy JC. Intestinal anastomotic injury alters spatially defined microbiome composition and function. Microbiome. 2014 Sep 15;2:35. doi: 10.1186/2049-2618-2-35. eCollection 2014. PMID 25250176
- [Result] Nalluri-Butz H, Bobel MC, Nugent J, Boatman S, Emanuelson R, Melton-Meaux G, Madoff RD, Jahansouz C, Staley C, Gaertner WB. A pilot study demonstrating the impact of surgical bowel preparation on intestinal microbiota composition following colon and rectal surgery. Sci Rep. 2022 Jun 22;12(1):10559. doi: 10.1038/s41598-022-14819-1. PMID 35732882
- [Result] Williamson AJ, Jacobson R, van Praagh JB, Gaines S, Koo HY, Lee B, Chan WC, Weichselbaum R, Alverdy JC, Zaborina O, Shogan BD. Enterococcus faecalis promotes a migratory and invasive phenotype in colon cancer cells. Neoplasia. 2022 May;27:100787. doi: 10.1016/j.neo.2022.100787. Epub 2022 Mar 30. PMID 35366466
- [Result] Yu T, Guo F, Yu Y, Sun T, Ma D, Han J, Qian Y, Kryczek I, Sun D, Nagarsheth N, Chen Y, Chen H, Hong J, Zou W, Fang JY. Fusobacterium nucleatum Promotes Chemoresistance to Colorectal Cancer by Modulating Autophagy. Cell. 2017 Jul 27;170(3):548-563.e16. doi: 10.1016/j.cell.2017.07.008. PMID 28753429
- [Result] Agnes A, Puccioni C, D'Ugo D, Gasbarrini A, Biondi A, Persiani R. The gut microbiota and colorectal surgery outcomes: facts or hype? A narrative review. BMC Surg. 2021 Feb 12;21(1):83. doi: 10.1186/s12893-021-01087-5. PMID 33579260
- [Result] Besselink MG, van Santvoort HC, Buskens E, Boermeester MA, van Goor H, Timmerman HM, Nieuwenhuijs VB, Bollen TL, van Ramshorst B, Witteman BJ, Rosman C, Ploeg RJ, Brink MA, Schaapherder AF, Dejong CH, Wahab PJ, van Laarhoven CJ, van der Harst E, van Eijck CH, Cuesta MA, Akkermans LM, Gooszen HG; Dutch Acute Pancreatitis Study Group. Probiotic prophylaxis in predicted severe acute pancreatitis: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Feb 23;371(9613):651-659. doi: 10.1016/S0140-6736(08)60207-X. Epub 2008 Feb 14. PMID 18279948
- [Result] Nataraj BH, Ali SA, Behare PV, Yadav H. Postbiotics-parabiotics: the new horizons in microbial biotherapy and functional foods. Microb Cell Fact. 2020 Aug 20;19(1):168. doi: 10.1186/s12934-020-01426-w. PMID 32819443
- [Result] D'Auria E, Panelli S, Lunardon L, Pajoro M, Paradiso L, Beretta S, Loretelli C, Tosi D, Perini M, Bedogni G, Abdelsalam A, Fiorina P, Bandi C, Zuccotti GV. Rice flour fermented with Lactobacillus paracasei CBA L74 in the treatment of atopic dermatitis in infants: A randomized, double- blind, placebo- controlled trial. Pharmacol Res. 2021 Jan;163:105284. doi: 10.1016/j.phrs.2020.105284. Epub 2020 Nov 4. PMID 33157233
- [Result] Nagpal R, Wang S, Ahmadi S, Hayes J, Gagliano J, Subashchandrabose S, Kitzman DW, Becton T, Read R, Yadav H. Human-origin probiotic cocktail increases short-chain fatty acid production via modulation of mice and human gut microbiome. Sci Rep. 2018 Aug 23;8(1):12649. doi: 10.1038/s41598-018-30114-4. PMID 30139941